CLINICAL TRIAL: NCT04787952
Title: Searching for the New Mechanisms That Activate Brow Fat Tissue
Brief Title: Insight Into New Brown Adipose Tissue Activators.
Status: Completed | Type: Observational
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Sponsor
Other Study IDs: UMB24/02/2021
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Adiposity; Metabolic Complication; Metabolic Disturbance; Healthy; Obesity; Diet Habit; Nutritional and Metabolic Diseases
Keywords: brown adipose tissue, obesity, diabetes type 2
MeSH Terms: conditions — Obesity; Feeding Behavior; Nutritional and Metabolic Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1= healthy subjects: Inclusion criteria to the group 1 (healthy males) N=20:
  1. BMI <25 kg/m2;
  2. RR<140/90mmHg;
  3. age 21-43 years
  4. fasting glycemia <100mg/dl; 2h-OGTT <140mg/dl;
  5. no chronic disease
  Interventions: Other: cold expossure
- Group 2 = overweight/obese subjects: Inclusion criteria to the group 2 ( overweight/obese males ) N=20:
  1. Blood pressure < 140/90 mmHg (well controlled by inh ACE; no beta-blockers)
  2. No chronic disease
  3. BMI > 25 <35kg/m²
  4. fasting glycemia <100mg/dl; 2h-OGTT <140mg/dl;
  5. age 21-43 years
  Interventions: Other: cold expossure

INTERVENTIONS:
Other: cold expossure — subjects were exposed for the cold, to activate and diagnose potential brown tissue activity

SUMMARY:
The general purpose of the study was to provide new information about the role of macronutrients intake, metabolomics, proteomics and microRNA on BAT activation.

The invesigator evaluated BAT activity and whole body energy consumption under cold stimulation in two gruops of healthy males aged 21-43 years old with normal BMI ( 19-25kg/m2) and in overweight/obese subjects.

DETAILED DESCRIPTION:
In detail, the main objectives of this study was to measure the influence of biological molecules of such fields: genomics, transcriptomics metabolomics and protemics and its relationship on BAT activation. The investigator also evaluated the role of diet, macronutirnets intake and polyunsaturated fatty acids on BAT activity.

Study design:

1. SCREENING VISIT:

* obtaining written informed consent from all subjects
* physical examination
* body composition analysis ( DXA + bioindepedance method inbody 720)

Laboratory analyses:

* Oral glucose tolerance test ( OGGT 75g)
* Morphology
* CRP
* Creatinine
* Urine analysis
* Lipids profile
* TSH
* ALT,AST

Dietary analysis All subjects fulfilled a 3-day food diary. Subjects were asked to compare the portion sizes with the colour photographs of each portion size, and to weigh food, if possible. The daily total energy, macronutrients, monounsaturated fatty acids (MUFA), polyunsaturated fatty acids (PUFA), omega-3, and omega-6 fatty acids intake were analysed.

2) STUDY VISITS: Patients who met the inclusion criteria and passed the screening stage were invited for the first visit when PET / MRI after 2h of cold exposure was performed.

Subjects were studied in the morning, from approximately 8 a.m. to 12 a.m., after an overnight fast beginning at 10 p.m. the night before. At the beginning of the day on which the PET study was performed, a catheter was inserted in the subject's antecubital vein for a bolus injection of 18F-FDG. Another catheter was inserted in the antecubital vein of the contralateral arm and was used to obtain samples of venous blood.

The subjects rested in a supine position under thermoneutral conditions (22°C) for 1 hour and then participants were exposed to cooling for 2 hours. The water perfused blankets were used in the applied protocol of cooling. Blood samples were taken before as well as in 60th and 120th min of cooling. Subjects were cooled until shivering and then temperature is set slightly (1-2°C) above the temperature that causes the onset of shivering. Shivering were confirmed by visual inspection and by asking the subject each 15 min. After 2 hour the tracer 18F-FDG (4 MBq/kg ) was administered intravenously, and scanning was performed after the injection of tracer.

Skin temperatures were measured continually by means of electrode attached to skin below armpit.

During the cold exposure, whole body resting energy expenditure (REE) was assessed by a computed open-circuit indirect calorimetry method- based on the consumption of O2 and the production of CO2. The 30 min long measurements of resting oxygen uptake and resting carbon dioxide production were performed by a ventilated canopy Vmax Encore 29n System (Viasys HealthCare, Yorba Linda, CA, USA) at the baseline ( -30 min to 0 min) and every 30 min until 120 min of cold exposure.

During PET-MRI scanning blood samples were taken in 5', 10' 20' 30' 40' to check the activity of 18-FDG. After PET/MRI patient's urine was collected and analyzed for activity of tracer. Blood samples were taken for analysis before the cold exposure, at 60 min and 120 min during the cold exposure to evaluate:

Glucose, IL-6, Insulin, Free Fatty Acids (FFA), TSH, fT4,fT3, Irisin, Atrial natriuretic peptide (ANP), Brain natriuretic peptide (BNP), plasma nonesterified fatty acid (NEFA), DNA, Peripheral Blood Mononuclear Cell (PBMC) for microRNA isolation, metabolomics and proteomics analysis.

SUMMARY:

The goal of our study is to search for new mechanisms that stimulate activation of BAT. It is likely that individuals with different content and activity of the brown adipose will have different set of serum markers after exposure to cold. This will allow the identification of new biomarkers and to understand the molecular mechanisms responsible for the activation of the brown adipose tissue. The outcomes will enable to find new potential therapeutic and diagnostic applications given to the current obesity pandemic.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria to the group 1 (healthy males) N=20:

1. BMI <25 kg/m2;
2. RR<140/90mmHg;
3. age 20-30/40 years
4. fasting glycemia <100mg/dl; 2h-OGTT <140mg/dl;
5. no chronic disease

Inclusion criteria to the group 2 ( overweight/obese males) N=20:

1. Blood pressure < 140/90 mmHg (well controlled by inh ACE; no beta-blockers)
2. No chronic disease
3. BMI > 25 <35kg/m²
4. fasting glycemia <100mg/dl; 2h-OGTT <140mg/dl;

Exclusion Criteria:

1. Any drug use: beta-blokers, statins, glucocorticoids drugs, hypertension drugs;
2. hypertension;
3. cancer;
4. hormonal disorders;
5. Inflammation process
6. Smoking
7. Claustrophobia

Ages: 20 Years to 43 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity.
Study Population: The study group comprised of 28 young, healthy, non - smoking Caucasian males, aged 21-42 years (mean age 26.75 ±5.11 years old), 16 with normal body weight (BMI < 25 kg/m2) and 12 obese/overweight (BMI > 25 kg/m2). Only participants without any comorbidities (e.g. hypo- and hyperthyroidis, asthma, cardiovascular disease, renal and liver failure, etc.) as well as without any medications (beta-blockers etc.) that could have impact on results, were enrolled to the study. Outside and shift workers have been excluded from the study as well.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2018-02-24 (Actual); Study Completion 2018-02-24 (Actual)

PRIMARY OUTCOMES:
The potential associations between BAT activity and dietary intake | 2016-2018
  The relationship between BAT activity and dietary intake will be analyzed
The potential associations between BAT activity and metabolite profile | the baseline (before cold exposure) and after 1st hour and 2nd hour of cold exposure
  The potential molecules will be identified by metabolomics approach and will be analyzed dependently on the brown tissue activity level
The potential associations between BAT activity and proteins profile | the baseline (before cold exposure) and after 1st hour and 2nd hour of cold exposure
  The potential molecules will be identified by proteomics approach and will be analyzed dependently on the brown tissue activity level
The potential associations between BAT activity and transcriptome profile | the baseline (before cold exposure) and after 1st hour and 2nd hour of cold exposure
  The potential molecules will be identified by transriptomics approach and will be analyzed dependently on the brown tissue activity level

SECONDARY OUTCOMES:
The potential associations between BAT activity and Interleukin-6 concentrations | the baseline (before cold exposure) and after 1st hour and 2nd hour of cold exposure
  The IL-6 concentration was measured before and during cold exposure and analyzed dependently on brown adipose tissue activity
The potential associations between BAT activity and energy expenditure | at the baseline ( -30 min to 0 min) and every 30 min until 120 min of cold exposure
  The energy expenditure was measured before and during the cold exposure, and analyzed dependently on brown adipose tissue activity
The potential associations between BAT activity and substrates utilization | at the baseline ( -30 min to 0 min) and every 30 min until 120 min of cold exposure.
  The substrates utilization was measured before and during the cold exposure, and analyzed dependently on brown adipose tissue activity
The potential associations between BAT activity and glucose concentrations | he baseline (before cold exposure) and after 1st hour and 2nd hour of cold exposure
  The glucose concentration was measured before and during cold exposure and analyzed dependently on brown adipose tissue activity
The potential associations between BAT activity and insulin concentrations | the baseline (before cold exposure) and after 1st hour and 2nd hour of cold exposure
  The insulin concentration was measured before and during cold exposure and analyzed dependently on brown adipose tissue activity
The potential associations between BAT activity and FFA ( free fatty acids) concentrations | the baseline (before cold exposure) and after 1st hour and 2nd hour of cold exposure
  The FFA concentration was measured before and during cold exposure and analyzed dependently on brown adipose tissue activity
The potential associations between BAT activity and irisin concentrations | the baseline (before cold exposure) and after 1st hour and 2nd hour of cold exposure
  The irisin concentration was measured before and during cold exposure and analyzed dependently on brown adipose tissue activity
The potential associations between BAT activity and atrial natiuretic peptide concentrations | the baseline (before cold exposure) and after 1st hour and 2nd hour of cold exposure
  The atrial natriuretic peptide concentration was measured before and during cold exposure and analyzed dependently on brown adipose tissue activity
The potential associations between BAT activity and brain natiuretic peptide concentrations | the baseline (before cold exposure) and after 1st hour and 2nd hour of cold exposure
  The brain natriuretic peptide concentration was measured before and during cold exposure and analyzed dependently on brown adipose tissue activity
The potential associations between BAT activity and plasma nonesterified fatty acid concentrations | the baseline (before cold exposure) and after 1st hour and 2nd hour of cold exposure
  The plasma nonesterified fatty acid concentration was measured before and during cold exposure and analyzed dependently on brown adipose tissue activity
The potential associations between BAT activity and TSH concentrations | the baseline (before cold exposure) and after 1st hour and 2nd hour of cold exposure
  The TSH concentration was measured before and during cold exposure and analyzed dependently on brown adipose tissue activity
The potential associations between BAT activity and fT3 concentrations | the baseline (before cold exposure) and after 1st hour and 2nd hour of cold exposure
  The fT3 concentration was measured before and during cold exposure and analyzed dependently on brown adipose tissue activity
The potential associations between BAT activity and fT4 concentrations | the baseline (before cold exposure) and after 1st hour and 2nd hour of cold exposu
  The fT4 concentration was measured before and during cold exposure and analyzed dependently on brown adipose tissue activity

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Maliszewska, PhD, Principal Investigator — Medical University of Bialystok, Poland

IPD SHARING:
Plan to Share IPD: Yes
Data maybe shared upon reasonable request and according with the Medical University of Bialystok condition.
Access Criteria: Data maybe shared upon reasonable request and according with the Medical University of Bialystok condition.